CLINICAL TRIAL: NCT03236948
Title: Individually Randomised Control Trial Evaluation of the Effectiveness of the Women for Women International (WfWI) Intervention in Afghanistan for Intimate Partner Violence Prevention Among Married Women
Brief Title: RCT of the Effectiveness of the WfWI Intervention in Afghanistan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: Women for Women International (WfWI) (Unknown)
Responsible Party: Principal Investigator, Rachel Jewkes, Director Gender and Health Research Unit, Medical Research Council, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC034-11-2015
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Domestic Violence; Depressive Symptoms; Livelihoods
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Individual level randomised trial, with intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WfWI Intervention (Experimental): Women receive the WfWI intervention. This comprises of three main components. First, a social empowerment and health intervention. Second a livelihood strengthening intervention, including numeracy training, and vocational training. Third, a cash transfer conditional on attendance at the intervention to cover costs of attendance and provide start-up capital. The intervention is delivered over 12 months.
  Interventions: Behavioral: Women for Women International Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Women for Women International Intervention
  Arms: WfWI Intervention

SUMMARY:
This is an individually randomised control trial to assess the effectiveness of a livelihoods and social empowerment intervention, delivered by Women for Women International, on married women's experiences of intimate partner violence in Afghanistan. It has a 22 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Women should be in the lowest economic level (earning less than US$1.25/day)
* Unemployed
* No in education/school
* Not involved in a similar programme
* Able to provide informed consent

Exclusion Criteria:

* Not mentally incapacitated, so as unable to provide informed consent
* Already been part of the WfWI intervention previously

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1461 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Any past year physical intimate partner violence experienced amongst currently married women | 22 months post baseline
  Physical intimate partner violence is assessed using five items based on the WHO VAW scale. A positive response to any item leads to a person being classified as experiencing in the past year.
Past year severe physical intimate partner violence experience amongst currently married women | 22 months post baseline
  Severe physical intimate partner violence experience is assessed using 5 items. Past year severe physical IPV is assessed as positive if a person responds to two (or more) items as once, or one item as few (or more), essentially creating a more than once categorization.
Depressive symptomology | 22 months post baseline
  Past week depressive symptomology is assessed by the Centre for Epidemiological Studies Depression (CESD) scale, with the full twenty items. A mean score will be calculated.

SECONDARY OUTCOMES:
Household food insecurity in past four weeks | 22 months post baseline
  Three items ask about household level food insecurity in the past 4 weeks. A mean score is calculated.
Financial shock resilience | 22 months post baseline
  One item assesses ability to mobilise cash in an emergency.
Monthly earnings | 22 months post baseline
  A single item assesses women's past month earnings
Total savings | 22 months post baseline
  A single item assesses women's total savings
Life satisfaction | 22 months post baseline
  Life satisfaction is assessed using four-items derived from the Satisfaction With Life Scale. A mean score is produced.
Suicidal ideation in past 4 weeks | 22 months post baseline
  A single item assesses thoughts about suicide in past week.
Gender attitudes | 22 months post baseline
  11 questions assess women's gender attitudes. A mean score is created.
Married women's participation in household decision-making | 22 months post baseline
  Five items are asked about women's ability to participate in household decisions. A mean score is created.
Any emotional abuse in the past year amongst currently married women | 22 months post baseline
  Seven items assess emotional abuse in the past year. A mean score is calculated.
Perceptions of husband cruelty amongst currently married women | 22 months post baseline
  Five items ask about married women's perceptions of her husband and his attitudes and relationship towards her. A mean score is created
Mother-in-law or abuse in the past 12 months amongst currently married women | 22 months post baseline
  A single item assesses whether mother-in-laws have hit the woman in the past 12 months and another item assesses whether siblings have hit the woman in the past 12 months, an affirmative response to either item would indicate abuse.
Perceptions of mother-in-law cruelty amongst currently married women | 22 months post baseline
  For married women, six items ask about their relationship and the mother-in-laws attitudes towards her

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jewkes, PhD, Principal Investigator — Director Gender and Health Research Unit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibbs A, Corboz J, Chirwa E, Mann C, Karim F, Shafiq M, Mecagni A, Maxwell-Jones C, Noble E, Jewkes R. The impacts of combined social and economic empowerment training on intimate partner violence, depression, gender norms and livelihoods among women: an individually randomised controlled trial and qualitative study in Afghanistan. BMJ Glob Health. 2020 Mar 16;5(3):e001946. doi: 10.1136/bmjgh-2019-001946. eCollection 2020. PMID 32201622
- [Derived] Gibbs A, Said N, Corboz J, Jewkes R. Factors associated with 'honour killing' in Afghanistan and the occupied Palestinian Territories: Two cross-sectional studies. PLoS One. 2019 Aug 8;14(8):e0219125. doi: 10.1371/journal.pone.0219125. eCollection 2019. PMID 31393873
- [Derived] Gibbs A, Corboz J, Jewkes R. Factors associated with recent intimate partner violence experience amongst currently married women in Afghanistan and health impacts of IPV: a cross sectional study. BMC Public Health. 2018 May 3;18(1):593. doi: 10.1186/s12889-018-5507-5. PMID 29724222
- [Derived] Gibbs A, Corboz J, Shafiq M, Marofi F, Mecagni A, Mann C, Karim F, Chirwa E, Maxwell-Jones C, Jewkes R. An individually randomized controlled trial to determine the effectiveness of the Women for Women International Programme in reducing intimate partner violence and strengthening livelihoods amongst women in Afghanistan: trial design, methods and baseline findings. BMC Public Health. 2018 Jan 22;18(1):164. doi: 10.1186/s12889-018-5029-1. PMID 29357843